CLINICAL TRIAL: NCT01920100
Title: Resource Use and Disease Course in Dementia (REDIC)
Acronym: REDIC
Status: Completed | Type: Observational
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Norwegian Directorate of Health (Other Government); King's College London (Other); Karolinska Institutet (Other); Oslo University Hospital (Other); University Hospital, Akershus (Other); Helse Midt-Norge (Other); Norwegian University of Science and Technology (Other); University of Bergen (Other); Norwegian Centre for Ageing and Health (Other)
Responsible Party: Sponsor
Other Study IDs: E13237
Record Dates: First submitted 2013-08-05; First posted 2013-08-09 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Neurodegenerative Diseases; Dementia
Keywords: Health Care Costs; Genetic Polymorphism
MeSH Terms: conditions — Neurodegenerative Diseases; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA samples are collected by mouth swabs from persons recruited from nursing homes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Memory clinic: People visiting a memory clinic at Ullevål University Hospital, St Olav Hospital or Innlandet Hospital Trust (n=400). The patients will be assessed three times over a three-year follow-up. Baseline inclusion started in January 2010. The final assessments will take place in spring 2014.
- Nursing homes: People admitted to a nursing home recruited from municipalities in Hedmark, Oppland, Nord-Trøndelag and Bergen (n=1000). Baseline assessments take place when the person is admitted to the nursing home. The patients will be assessed every six months over a three-year follow-up period. The first participant was included in March 2012, and baseline inclusion will be completed in December 2013.
- In-home care: People 70 years of age or older receiving in-home care recruited from municipalities in Hedmark, Oppland, Oslo, Østfold and Buskerud (n=995). The patients will be assessed three times over a three-year follow-up period. Baseline inclusion started in April 2009 and the final assessments will take place in December 2013.
- People without dementia: People without dementia recruited from Nord-Trøndelag, Drammen and Oslo (n=400).
  The participants will be assessed three times over a three-year follow-up period. Baseline inclusion will take place in autumn 2012 and the last follow-up will take place in autumn 2015.

SUMMARY:
This project is based on a three-year program that aims to improve the knowledge of the socioeconomic consequences of dementia in Norway. By including patients with and without dementia in four different cohorts (from nursing homes, from memory clinics, home-dwelling persons with dementia and elderly persons without dementia), the project's aim is to describe the course of dementia, the economical cost of dementia and to look into possible risk factors for dementia.

ELIGIBILITY:
Memory clinic sample

Inclusion Criteria:

* All patients examined at a memory clinic with mild cognitive impairment or mild dementia

Exclusion Criteria:

* None

In-home care sample

Inclusion Criteria:

* Persons 70 years of age or older receiving in-home care from the municipality

Exclusion Criteria:

* None

Nursing-home sample

Inclusion Criteria:

* All persons admitted to the nursing home with an expected stay of more than four weeks.
* Participants should be 65 years or older, unless established dementia disease, in which case younger persons also will be included

Exclusion Criteria:

* Life expectancy of less than six weeks

Control sample

Inclusion Criteria:

* Persons 65 years or older without any sign of dementia

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nursing home Memory clinics In-home care Persons without dementia (Control)
Sampling Method: Non-Probability Sample
Enrollment: 696 (Actual)
Dates: Start 2009-04; Primary Completion 2015-01 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
Cost of dementia | 3 years
  The cost of dementia is assessed with the Resource Utilization in Dementia (RUD) (Wimo et al. 2009), for a period of three years for all the four cohorts. The nursing home cohort is assessed at baseline and every 6 month for three years, the other three cohorts are assessed three times over a three-year follow up period.

SECONDARY OUTCOMES:
The course of neuropsychiatric symptoms | 3 years
  The course of neuropsychiatric symptoms (depression, anxiety, psychosis, aggression, apathy, and cognition, are assessed with standardized assessment Tools. The nursing home cohort is assessed at baseline and every 6 month for three years, the other three cohorts are assessed three times over a three-year follow up period.
Quality of Life in persons admitted to nursing homes | 3 years
  Quality of Life is assessed with standardized assessment Tools. The nursing home cohort is assessed at baseline and every 6 month for three years, the other three cohorts are assessed three times over a three-year follow up period.
Prescription of medication | 3 years
  Prescription of medication is recorded at baseline, and the amount of medication used is recorded throughout the study period. The nursing home cohort is assessed at baseline and every 6 month for three years, the other three cohorts are assessed three times over a three-year follow up period.
DNA polymorphism | At baseline
  DNA samples are collected for the nursing home cohort, and they are assessed for genetic polymorphism previous associated with dementia. The results are used as covariates in the analyses of the course of the symptoms and to look for risk factors for dementia.
Organizational factors of the nursing homes | At baseline
  Organizational factors of the nursing homes and variables associated with the staff of the nursing homes will be collected at baseline, and the data will be used to explore associations between nursing home characteristics and the course of the symptoms in the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Geir Selbaek, pHd, Principal Investigator — Centre for old age psychiatry research, Innlandet Hospital Trust
Locations (3):
- Norway (3):
  - University of Bergen, Bergen
  - Senter for omsorgsforskning - Midt, Namsos
  - Innlandet Hospital Trust, Ottestad

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Sandvik RKNM, Husebo BS, Selbaek G, Strand G, Patrascu M, Mustafa M, Bergh S. Oral symptoms in dying nursing home patients. Results from the prospective REDIC study. BMC Oral Health. 2024 Jan 25;24(1):129. doi: 10.1186/s12903-024-03901-x. PMID 38273300
- [Derived] Callegari E, Saltyte Benth J, Selbaek G, Gronnerod C, Bergh S. Do prescription rates of psychotropic drugs change over three years from nursing home admission? BMC Geriatr. 2021 Sep 16;21(1):496. doi: 10.1186/s12877-021-02437-x. PMID 34530728
- [Derived] Sandvik RK, Selbaek G, Bergh S, Aarsland D, Husebo BS. Signs of Imminent Dying and Change in Symptom Intensity During Pharmacological Treatment in Dying Nursing Home Patients: A Prospective Trajectory Study. J Am Med Dir Assoc. 2016 Sep 1;17(9):821-7. doi: 10.1016/j.jamda.2016.05.006. Epub 2016 Jun 16. PMID 27321869
- See also: Link to web page with a working paper describing the project — http://www.med.uio.no/helsam/english/research/publications/working-papers/heled/2012/redic.html